CLINICAL TRIAL: NCT00709046
Title: High Dose Versus Standard Dose Proton Pump Inhibitor in High-risk Bleeding Peptic Ulcers After Combined Endoscopic Hemostasis: A Prospective Randomized Comparative Study
Brief Title: High Dose Versus Standard Dose Proton Pump Inhibitor (PPI) in High-risk Bleeding Peptic Ulcers After Combined Endoscopic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chieh-Chang Chen, National Taiwan Univeritsy Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200710033M
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Endoscopy; Peptic Ulcer; Bleeding; Proton Pump Inhibitors
Keywords: Endoscopic treatment; Peptic ulcer; Bleeding; Thermocoagulation; Proton pump inhibitors
MeSH Terms: conditions — Peptic Ulcer; Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): High dose pantoprazole infusion
  Interventions: Drug: High dose pantoprazole infusion
- 2 (Active Comparator): standard dose pantoprazole infusion
  Interventions: Drug: Standard dose pantoprazole infusion

INTERVENTIONS:
Drug: High dose pantoprazole infusion — Pantoprazole 80mg iv bolus, 8mg/hr infusion for 72hrs
  Other Names: Pantoloc
  Arms: 1
Drug: Standard dose pantoprazole infusion — Pantoprazole 40mg iv bolus qd x 3 days
  Other Names: Pantoloc
  Arms: 2

SUMMARY:
The study was designed to evaluate the efficacy an adjuvant use of standard dose or high dose of proton pump inhibitor after combined endoscopic hemostasis therapy.

DETAILED DESCRIPTION:
Acute peptic ulcer bleeding remains the most common cause of acute upper gastrointestinal bleeding. Endoscopy serves as a tool for initial diagnosis and triage and also a tool for immediate hemostasis, especially for high-risk lesions. High-risk lesions include peptic ulcers with active spurting vessel, oozing vessel, or NBVV, nonbleeding visible vessel. Current modalities of endoscopic hemostasis include epinephrine injection, endoscopic coaptive thermocoagulation, hemoclipping. Endoscopic hemostasis has been documented by a number of clinical studies to be effective in decreasing rebleeding, need for emergency surgery, decreasing hospitalization days. Current evidence also shows that combination therapy with epinephrine injection and heater probe thermocoagulation/hemo-clip hemostasis is more effective than epinephrine injection alone or than heater probe thermocoagulation alone, or than hemoclip hemostasis alone. Studies showed a high dose intravenous proton pump inhibitor infusion after initial endoscopic hemostasis reduced recurrent ulcer bleeding. However, it was still controversial whether an adjuvant use of standard-dose proton pump inhibitor therapy to endoscopic therapy had similar benefit. We hypothesized that an adjuvant use of standard dose of proton pump inhibitor after combined endoscopic hemostasis therapy offer similar benefit as high dose proton pump inhibitor did.

ELIGIBILITY:
Inclusion Criteria:

* adults aged above 16 years old with acute nonvariceal upper gastrointestinal bleeding
* read, agree to attend the study, and signed informed consent indicated to receive esophagogastroduodenoscopy(EGD)
* peptic ulcers with high risk lesions (active bleeding: spurting, oozing peptic ulcers. Ulcers with NBVV: nonbleeding visible vessel)

Exclusion Criteria:

* unable to receive EGD (unable to open mouth, upper gastrointestinal obstruction)
* bleeding tendency (platelet < 50x109/L, prothrombin time INR >2, ongoing use of heparin or coumadin)
* gastric malignancy
* myocardial infarction within recent one week
* recent cerebrovascular event within recent one week
* pregnancy
* refuse to attend the study
* known allergy history to epinephrine or pantoprazole

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
rate of initial hemostasis and the rate of recurrent bleeding | 72hr

SECONDARY OUTCOMES:
need for surgical intervention to control bleeding, transfusion requirements, length of hospital stay (in days), and 30-day mortality | 30day

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen CC, Lee JY, Fang YJ, Hsu SJ, Han ML, Tseng PH, Liou JM, Hu FC, Lin TL, Wu MS, Wang HP, Lin JT. Randomised clinical trial: high-dose vs. standard-dose proton pump inhibitors for the prevention of recurrent haemorrhage after combined endoscopic haemostasis of bleeding peptic ulcers. Aliment Pharmacol Ther. 2012 Apr;35(8):894-903. doi: 10.1111/j.1365-2036.2012.05047.x. Epub 2012 Feb 28. PMID 22369682